CLINICAL TRIAL: NCT00549250
Title: Human Papillomavirus 6/11 in the Lower Airway of Neonates
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 200710007R
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-06

CONDITIONS: Papillomavirus Infections
Keywords: Human papillomavirus 6/11; Neonates; Human papillomavirus 6 or 11 infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bronchial lavage fluid
Oversight: Data Monitoring Committee: No

SUMMARY:
Vertical transmission of human papillomavirus (HPV) 6/11 leads to infection in the lower airway of neonates. The presence of HPV 6/11 may later cause juvenile onset recurrent respiratory papillomatosis (JORRP).

DETAILED DESCRIPTION:
Juvenile onset recurrent respiratory papillomatosis (JORRP) is caused by human papillomavirus (HPV), almost exclusively type 6 and 11. The disease is well-known for its recurrence and difficulty in management. The peak incidence is around 2-3 year of age. Since HPV infection has always been considered a sexual transmitted disease, the rate of vertical or perinatal transmission had been studied extensively. However, few studies focused on HPV 6 and 11.

To the best of our knowledge, in the several large-scale studies available for HPV infection in the newborn, no case of HPV 6/11 infection had been identified. Most of these studies had specimens taken from the oral cavity of newborn. In contrast to the occurrence of JORRP in the larynx, trachea and lower respiratory tract, if vertical transmission of HPV 6/11 does exist, specimens from lower respiratory tract of newborn is mandatory to detect any possible infection.

There is no study available about HPV 6/11 infection in the lower airway of healthy neonate/children. In some studies of adults, the prevalence of HPV 6/11 in larynx or vocal cord of patients without recurrent respiratory papillomatosis ranged between 19~25%. In contrast, several studies had specimen taken from the non-disease lower airway (trachea, vocal cord) and/or larynx of patients with JORRP. Except for the almost 100% presence of HPV 6/11 DNA in the diseased site, 38~60% of specimens taken from non-disease site were also positive for the viral DNA, showing that latent infection is not infrequent in normal airway, and may later cause active disease by mechanism still unknown to date.

The largest national registry of JORRP to date was conducted in the US and had 603 cases. The study showed that there was a significant association between younger age at diagnosis and papillomas occurring below the larynx (mean age 4.6 VS 2.1 years, p=0.009). This finding further emphasizes the importance of getting specimen at the laryngeal level, especially in neonates.

The aim of our study is to examine the presence of HPV 6/11 DNA in lower respiratory tract specimens from newborn. To get the lower respiratory tract specimen without unnecessary medical intervention, only those needed intubation will be included in this study. Specimens from bronchial lavage (or scraping?) will be obtained after getting informed consent from the parents, and undergo PCR to identify the presence of HPV 6/11 DNA.

ELIGIBILITY:
Inclusion Criteria:

* In order to get respiratory specimens at or below the larynx, intubated neonates younger than one-month-old admitted to our neonatal intensive care unit will be included in this study after getting informed consent from their families.

Exclusion Criteria:

* Unless the neonate's condition is too critical to have the following procedure performed, gestational age, co-morbidity and maternal status of HPV infection are not exclusion criteria for this study.

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All intubated neonates younger than 1 month-old admitted to our neonatal intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is to identify prospectively the presence and the estimated prevalence of HPV 6/11 DNA in the lower airway of neonates by polymerase chain reaction (PCR). | sampling time

CONTACTS AND LOCATIONS:
Overall Officials: Li-Min Huang, M.D.Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan